CLINICAL TRIAL: NCT04169477
Title: Superiority, Prospective, Multicentric, Randomized, Single-blind, Cross-over Study Comparing 2 Modes of Transcutaneous Electrical Nerve Stimulation (TENS) in Chronic Neuropathic Radiculalgia
Brief Title: Comparison of Two Modes of Transcutaneous Electrical Nerve Stimulation (TENS) in Chronic Neuropathic Radiculalgia
Acronym: CROSS-TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RC-P0080; 2018-A03074-51 ID RCB (Other: ANSM France)
Record Dates: First submitted 2019-11-05; First posted 2019-11-20 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Neuropathic Pain; Radiculopathy
Keywords: TENS
MeSH Terms: conditions — Neuralgia; Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTENS-mTENS (Experimental): Patients randomized in this arm will test cTENS mode first, the subjects will be crossed over to the mTENS form
  Interventions: Device: CEFAR Primo Pro (TENS device)
- mTENS-cTENS (Experimental): Patients randomized in this arm will test mTENS mode first, the subjects will be cross over to the cTENS mode
  Interventions: Device: CEFAR Primo Pro (TENS device)

INTERVENTIONS:
Device: CEFAR Primo Pro (TENS device) — During the first month: Patients will have to test 3 sessions of TENS 1 hour/day. Depending on their arm assigned by randomization, patients will begin with c-TENS or m-TENS.
  [Cross-over] During the second month: Patients will test the other type they do not have used yet according to the following scheme: 3 sessions of 1 hour, each day.
  In this way, all patients will test successively the 2 different modes. After the end of the second month and up to the end of their participation (6 months after randomization) patients will be free to use the mode of TENS they prefer.

SUMMARY:
This study will compare 2 types of Transcutaneous Electrical Nerve Stimulation (TENS) to treat chronic neuropathic pain. TENS involves the application of electrical stimulation to the skin via surface electrodes to stimulate nerve fibres for pain relief.

DETAILED DESCRIPTION:
TENS is already recommended in clinical practice to treat chronic neuropathic pain. The objective of this study is to compare the efficacy of 2 different modes of TENS: conventional TENS (c-TENS) and mixed-frequency TENS (m-TENS). Randomization will determine the mode that the patient has to test during the first month.

Each patient will test successively each mode during 1 month at home (3 sessions 1 hour/day). Then, the patient will test the other mode during the second month. Up to 6 months, the patient will be free to use the mode of TENS he wants.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or older
* Patients with chronic neuropathic radiculalgia from at least 3 months of evolution
* Radiculalgia VAS > or egal to 40/100
* Neuropathic pain diagnostic (DN4) score > or egal to 4
* Patient who has accepted to participate in the study by signing the informed consent form

Exclusion Criteria:

* Pregnancy
* Dermatosis in the painful dermatome
* Venous or arterial thrombosis of the lower limbs
* Patient with active implantable medical device
* Severe cognitive disorders
* Patient under a legal protection regime(guardianship/curatorship/guardianship of justice)
* Previous use of TENS to treat radiculalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Change in the visual analog scale for evaluation of radiculalgia (from 0 to 100) | day 30, day 60
  Visual analogue scales are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain being 0 equivalent to no pain and 100 to the worst possible pain

SECONDARY OUTCOMES:
Patient preference rate | day 60
  After having tested each mode during one month, the patients will be asked to give their preference (c-TENS or m-TENS)
Patient Global Impression of Change (PGIC) | day 30, day 60
  Patient Global Impression of Change is a 7-point scale used by the patient to rate the severity of the patient's illness at the time of assessment being 1 equivalent to no change or worsening and 7 to very much improved, making a difference
Rate of patient compliance | day 30, day 60
  Rate of TENS sessions completed by the patient compared to the number of sessions prescribed for each mode
Rate of patients with adverse events | day 30, day 60, day 180
  Rate of patients with adverse events definitely or possibly attributable to neurostimulation for each type
Brief pain inventory (impact on daily life) (BPI) | day 30, day 60
  The BPI allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. There are line drawings of the front and back of a human body on which patients mark the location of their pain. In addition, patients fill out 11 different questions about pain intensity (present as well as least, most, and average for the past 24 hours) and the effect of the pain on their ability to function during various activities of daily living (pain interference items) rated on 0-10 scales being equivalent to no interference and 10 to complete interference.
Mean of post-effect delay | day 60
  for each mode of TENS, patient estimation between end of a TENS session and return to initial intensity of the pain (calculated from patient journal completed every day during the 2 first months of the study
Visual analog scale for evaluation of radiculalgia one month after | day 30, day 60
  Visual analogue scales are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain being 0 equivalent to no pain and 100 to the worst possible pain
Visual analog scale for evaluation of radiculalgia six months after | day 180
  Visual analogue scales are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain being 0 equivalent to no pain and 100 to the worst possible pain
Rate of therapeutic persistence according toTENS mode | day 180

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ducoulombier, MD, Principal Investigator — GHICL
Locations (4):
- France (4):
  - CH Béthune, Béthune
  - CHU Lille, Lille
  - GHICL, Lomme
  - CH Roubaix, Roubaix